CLINICAL TRIAL: NCT00543842
Title: Phase I/II Trial of Preoperative Radiotherapy With Concurrent Bevacizumab, Erlotinib and Capecitabine for Locally Advanced Rectal Cancer
Brief Title: Bevacizumab, Erlotinib, and Capecitabine for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0080
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Bevacizumab; Erlotinib; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Erlotinib Hydrochloride; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Erlotinib + Capecitabine + Radiation Therapy (Experimental): Bevacizumab 5 mg/kg intravenous (IV) every 2 weeks for 3 Doses (Weeks 1, 3, 5). Erlotinib starting dose 50 mg orally daily Weeks 1-3. Capecitabine starting dose 650 mg/m^2 orally twice daily Monday-Friday for 6 Weeks. Radiation Therapy 30 minute radiation treatments, dose of 50.4 Gy once daily on 5 consecutive days, for up to 5 weeks and 3 days, totaling 28 treatments. At least 8 weeks after radiation therapy, surgical removal of rectal tumor.
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Erlotinib; Radiation: Radiation Therapy; Procedure: Surgery

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg By Vein Every 2 Weeks x 3 Doses (Weeks 1, 3, 5)
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Capecitabine — Starting Dose 650 mg/m^2 By Mouth Twice Daily Monday-Friday x 6 Weeks
  Other Names: Xeloda
Drug: Erlotinib — Starting Dose 50 mg By Mouth Daily Weeks 1-3
  Other Names: Erlotinib Hydrocloride; OSI-774; Tarceva
Radiation: Radiation Therapy — 30 minute radiation treatments, dose of 50.4 Gy once daily on 5 consecutive days, for up to 5 weeks and 3 days, totaling 28 treatments
  Other Names: RT; XRT; Radiotherapy
Procedure: Surgery — At least 8 weeks after radiation therapy, surgical removal of rectal tumor

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of bevacizumab (Avastin) and erlotinib hydrochloride (Tarceva) that can be given in combination with standard radiation therapy and capecitabine before surgery to patients with rectal cancer. The safety and effectiveness of this combination of therapies will also be studied.

The goal of this Phase I trial was to determine the maximal tolerated dose (MTD) of concurrent capecitabine, bevacizumab and erlotinib with preoperative radiation therapy (RT) for rectal cancer. The trial completed as Phase I without progressing to the Phase II portion.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Erlotinib hydrochloride is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Capecitabine is designed to interfere with the growth of cancer cells.

Study Phases:

The study has 2 parts, called Phase I and Phase II. In the Phase I portion, participants will be treated with 1 of 4 dose combinations of capecitabine, bevacizumab, and erlotinib hydrochloride, along with radiation therapy. The dose level of capecitabine and erlotinib hydrochloride will change during Phase I, but the dose levels of bevacizumab and radiation therapy is the same for all participants. The first group of participants will be given the lowest dose combination. If that group does not experience intolerable side effects, the next group of participants will be enrolled at a higher dose level. This will continue until the highest tolerable dose level of the study drug and radiation therapy combination is found (called the maximum tolerated dose, or MTD).

Based on the results of Phase I, researchers will decide the MTD level of chemotherapy and radiation therapy. In Phase II, participants will be treated at the MTD dose level. Up to 26 participants will be treated in each phase.

Radiation and Chemotherapy Administration:

If you are found to be eligible to take part in this study, you will begin radiation therapy. The radiation therapy will be given once a day for 5 days in a row (Monday-Friday) each week, for up to 5 weeks and 3 days. You will have up to a total of 28 radiation treatments. Each radiation treatment will take about 30 minutes.

You will take the chemotherapy drug capecitabine by mouth twice a day as a tablet on each of the days that you receive radiation therapy. These pills will not be taken on Saturday and Sunday. You must not be taking the drug cimetidine, and must be off of coumadin for at least 1 week and sorivudine and brivudine for at least 4 weeks before starting capecitabine and during the entire capecitabine therapy. If you are not able to stop taking coumadin, you will need extra blood tests performed throughout the study to check your bleeding and clotting speed.

You will receive the drug bevacizumab by vein once every 2 weeks for 6 weeks (a total of 3 doses). The infusion will at first last 90 minutes. If there are no allergic reactions, fevers, or chills after the first infusion, the infusion time for the second dose will be shortened to 60 minutes. If there is no allergic reactions or side effects during the second drug infusion, the last infusion of bevacizumab will be given over 30 minutes. If you do have some reactions to the infusion, you may receive extra preventive medications before the infusion, and the length of time may need to stay at 90 minutes.

You will take the chemotherapy drug erlotinib hydrochloride by mouth as a tablet once a day. Your doctor will tell you whether you will take erlotinib hydrochloride during the first 3 weeks of radiation therapy only, or during the whole time you are getting radiation therapy, up to 6 weeks.

Study Tests

During the study, you will have the following tests performed:

* You will have physical exams once a week.
* Every week, blood (about 2 teaspoons) will be drawn for routine tests.
* You will have a routine urine test in the first and third week of radiation therapy.
* The possible development of side effects will be closely monitored during weekly visits with your doctors.

At 6-8 weeks after you have stopped receiving radiotherapy, you will have a physical exam, routine blood tests (about 2 teaspoons), and a urine test.

Surgery:

At least 8 weeks after you have stopped receiving radiotherapy, you will have the rectal tumor removed by surgery. This is considered the standard of care and you will sign a separate surgical consent document.

Length of Study:

You will receive radiation therapy with capecitabine, bevacizumab, and erlotinib hydrochloride for 5 ½ to 6 weeks. At least 8 weeks after you stop receiving radiotherapy, you will have surgery. You may then receive additional chemotherapy.

You may be taken off study if the disease gets worse or you experience intolerable side effects.

Follow-up Testing:

After surgery and possible chemotherapy after surgery, you will be seen by a doctor every 3-4 months for 1 year, and then every 6 months for the next 3 years. You will have blood tests at these doctor visits. You will also have CT scans within 4-6 months after completion of chemotherapy then every 6 months for the first 3 years, and then once a year for the next 2 years. These tests are all the standard of care procedures for treatment of colorectal cancer.

This is an investigational study. Capecitabine and bevacizumab have been approved by the FDA for the treatment of metastatic colorectal cancer. Erlotinib hydrochloride has been approved by the FDA for treatment of pancreatic cancer, but not for colorectal cancer. The combination of capecitabine, erlotinib and bevacizumab with radiation therapy has not been approved by the FDA. At this time, this combination is being used in research only.

Update: Nineteen participants were enrolled at MD Anderson for the Phase I portion of the study then the study was completed December 2013.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
2. Patients must be >/= 18 years of age.
3. All patients must have histologically confirmed adenocarcinoma of the rectum with pathologic material reviewed by the Department of Pathology at MD Anderson Cancer Center (MDACC).
4. Patients must have clinical stage II-III (T3, T4 or node-positive) based on computed tomography (CT), magnetic resonance (MR) or endoscopic ultrasound criteria.
5. Patients must have no distant metastatic disease on chest, abdomen and pelvic CT scan performed with IV contrast. If the CT was performed outside of MDACC, the slice thickness must be </= 7.5 mm. Criteria for pathologic enlargement of lymph nodes is > 15 mm on short axis dimension.
6. The rectal tumor must be either palpable on digital rectal exam or the inferior edge of the tumor must be within 12 cm of the anal verge based on rigid proctoscopy.
7. Patients must have absolute neutrophil count (ANC) >/= 1500/L, platelets >/= 100,000/mm^3, total serum bilirubin less than 2.0 mg%, blood urea nitrogen (BUN) </= 30 mg%, creatinine </= 1.5 mg% and creatinine clearance >/= 30ml/min (estimated as calculated with Cockcroft-Gault equation). Note: In patients with moderate renal impairment (estimated creatinine clearance 30-50 mL/min) at baseline, a dose reduction to 75% of the capecitabine starting dose is recommended.
8. Hemoglobin >/= 9 gm/dL (may be transfused to maintain or exceed this level).
9. Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary. Patients must be made aware of their other treatment options.

Exclusion Criteria:

1. Prior radiotherapy to the pelvis.
2. Any prior chemotherapy.
3. Prior vascular endothelial growth factor (VEGF) or epidermal growth factor receptor (EGFR)-directed therapy, such as bevacizumab, cetuximab, erlotinib, or gefitinib.
4. Current, prior or planned participation in any other experimental drug study.
5. Pregnant or lactating woman. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Women / men of childbearing potential not using a reliable contraceptive method (oral contraceptive, other hormonal contraceptive, intrauterine device, diaphragm or condom). (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients must agree to continue contraception for 30 days from the date of the last study drug administration.
6. Serious, uncontrolled, concurrent infection(s) requiring intravenous (IV) antibiotics.
7. Treatment for other clinically significant cancers within the last five years, except cured non-melanoma skin cancer and treated in-situ cervical cancer.
8. Inadequately controlled hypertension [systolic blood pressure of >130 and/or diastolic blood pressure of >90 mmHg on antihypertensive medication at time of study entry and/or at time of starting therapy] history of myocardial infarction or unstable angina within 12 months prior to study enrollment, New York Heart Association Class II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible) or Class II or greater peripheral vascular disease
9. History of stroke or transient ischemic attack at any time,history of hypertensive crisis or hypertensive encephalopathy.
10. Aspartate aminotransferase or alanine aminotransferase (AST or ALT) >/= 2.5 times the upper limit of normal.
11. Inability to swallow oral medication.
12. Evidence of bleeding diathesis or coagulopathy, international normalized ratio (INR) >/= 2.5.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day 0.
14. Proteinuria at baseline or clinically significant impairment of renal function as demonstrated by either a. Urine protein:creatinine ratio >/= 1.0 at screening. b. Urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
15. Current serious, nonhealing wound, ulcer, or bone fracture.
16. History of aortic aneurysm > 4.5 or aortic dissection.
17. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
18. Patients who have had an organ allograft.
19. Patients on Coumadin are recommended to be changed to Low Molecular Weight Heparin (LMWH) at least 1 week prior to starting capecitabine. If patients cannot be switched to LMWH, then extra monitoring of their International Normalized Ratio (INR) will be performed.
20. Patients taking Sorivudine or Brivudine must be off of these drugs for 4 weeks. Patients taking cimetidine must have this drug discontinued. Ranitidine or a drug from another anti-ulcer class can be substituted for cimetidine if necessary. If patient is currently receiving allopurinol, must discuss with PI to see of another agent may substitute for it.
21. Patients with known Gilberts disease will be considered ineligible due to potential UGTA1 polymorphism effects on metabolism for erlotinib.
22. Inability to comply with study and/or follow-up procedures.
23. Known hypersensitivity to any component of bevacizumab, erlotinib or capecitabine
24. Prior history of hypertensive crisis or hypertensive encephalopathy
25. Peripheral arterial thrombosis within 6 months prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | Continuoual Reassessment Weeks 1- 6
  MTD derived from differing dose combinations of Capecitabine, Bevacizumab, and Erlotinib of using the continual reassessment method (CRM). Dose limiting toxicity defined as any grade 3 or higher acute toxicity during chemoradiation. The MTD will be defined as the dose at which grade 3 or higher acute toxicity exceeds 25%.

CONTACTS AND LOCATIONS:
Overall Officials: Prajnan Das, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org